CLINICAL TRIAL: NCT03546985
Title: A Randomized, Multi-center, Single-use, Active-controlled, Open Study to Assess the Local Analgesic Effect of Episil® Oral Liquid in Cancer Patients Suffering From Chemotherapy- and/or Radiation-induced Oral Mucositis
Brief Title: A Trial of Episil® Oral Liquid in Cancer Patients Suffering From Chemotherapy- and/or Radiation-induced Oral Mucositis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Solasia Pharma K.K. (Industry)
Collaborators: Solasia Medical Information Consulting (Shanghai) Co. Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SP-0301
Record Dates: First submitted 2018-04-23; First posted 2018-06-06 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2018-06

CONDITIONS: Chemotherapy- and/or Radiation-induced Oral Mucositis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental)
  Interventions: Device: episil®
- Group B (Active Comparator)
  Interventions: Device: Kang Su

INTERVENTIONS:
Device: episil® — Firmly press the pump and apply the stream of liquid to the oral cavity 3 times (a total volume of 0.45 mL approximately). Distribute to affected areas in the mouth, for example by using the tongue. Wait for 5 minutes for the protective film to form.
  Arms: Group A
Device: Kang Su — Gently pour 5 mL of rinse into the mouth, keep the rinse staying in the oral cavity for at least 1 minute, and spilt out the liquid.
  Other Names: Generic of MuGard®
  Arms: Group B

SUMMARY:
This is a randomized, multi-center, single-use, active-controlled, two-stage open study of episil®. The purpose of this study is to assess the local analgesic effect of episil® in cancer patients suffering from chemotherapy- and/or radiation-induced oral mucositis, which will provide scientific and reliable clinical data in the product registration in China.

ELIGIBILITY:
Inclusion Criteria:

* Male/female patient 18 years of age;
* Pathological histologic and/or cytological diagnosis of malignant tumor;
* Patients who are suffering from symptomatic oral mucositis (WHO grade 2 or above) during chemotherapy and/or radiotherapy during screening period;
* Patients who are suffering from pain inside the oral cavity caused by oral mucositis, and pain assessment by Likert scale (0-10) results in a score of at least 6 out of 10 during screening period and at enrollment on Day 1;
* Patients undergoing chemotherapy and/or radiotherapy: patients must have received at least one cycle of multiple-cycle chemotherapy regimen and/or have received multiple doses of radiation, prior to the enrollment on Day 1;
* Patients at Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, 2 and 3; and
* Patients are able to provide written informed consent to participate in the study freely after the nature of the study and disclosure of data has been explained to the patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-12-26 (Actual); Primary Completion 2018-05-08 (Actual); Study Completion 2018-05-25 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) of pain score of oral mucositis | During 6 hours after a single use of investigational medical device
  Oral mucosal pain is assessed by a numerical score (0-10 Likert-pain scale).

SECONDARY OUTCOMES:
Pain intensity decrease inside the oral cavity | During 6 hours after a single use of investigational medical device
  Oral mucosal pain is assessed by a numerical score (0-10 Likert-pain scale).
Peak pain intensity difference inside the oral cavity | During 6 hours after a single use of investigational medical device
  Oral mucosal pain is assessed by a numerical score (0-10 Likert-pain scale).
Incidence of adverse events | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Xinchen Sun, Principal Investigator — Jiangsu People's Hospital; Guoyao Tang, Principal Investigator — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University School of Medicine
Locations (7):
- China (7):
  - The People's Liberation Army 307 Hospital, Beijing, Beijing Municipality
  - Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Tongji Hospital, Wuhan, Hubei
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The People's Liberation Army 81 Hospital, Nanjing, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No